CLINICAL TRIAL: NCT03484858
Title: The Effects of Exercise on Glycaemic Response of Low or High Glycaemic Index Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015/01092
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Glycaemic Response
MeSH Terms: interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Randomized cross over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High glycaemic index meal and exercise (Other)
  Interventions: Other: High glycaemic index meal and exercise
- High glycaemic index meal and rest (Other)
  Interventions: Other: High glycaemic index meal and rest
- Low glycaemic index meal and exercise (Other)
  Interventions: Other: Low glycaemic index meal and exercise
- Low glycaemic index meal and rest (Other)
  Interventions: Other: Low glycaemic index meal and rest

INTERVENTIONS:
Other: High glycaemic index meal and exercise
  Arms: High glycaemic index meal and exercise
Other: High glycaemic index meal and rest
  Arms: High glycaemic index meal and rest
Other: Low glycaemic index meal and exercise
  Arms: Low glycaemic index meal and exercise
Other: Low glycaemic index meal and rest
  Arms: Low glycaemic index meal and rest

SUMMARY:
The aim of the current study is to determine the effect of sprint interval training (SIT) in conjunction with either high or low glycaemic index meals (breakfast, lunch and dinner) on the 24-hour glycaemic profile and glucoregulatory hormones in Asian males.

DETAILED DESCRIPTION:
The study will recruit 20 young healthy Asian men of Chinese descent. Subjects will visit our Clinical Nutrition Research Centre (CNRC) on 5 occasions: once for consenting, screening and familiarization with the exercise and testing equipment (screening), and four additional times, interspaced by a minimum of 3 days, to undergo a total of four study conditions. The four study trials combine SIT or rest and low or high GI diet in a 2 x 2 design, and will be assigned in randomized order: (RL) Rest and low GI, (SL) SIT and low GI, (RH) Rest and high GI, and (SH) SIT and high GI. The test conditions will have comparable foods with RL and SL diets comprising local foods of low glycaemic index and RH and SH diets comprising local foods of high glycaemic index. Randomization of study trials will be carried out using an online randomizer (www.randomizer.org/). In the SL and SH trials, subjects will perform a SIT bout consisting of alternating periods of low-resistance cycling (4 ½ minutes) and maximal effort all out cycling (30 sec Wingate test) for a total of 30 min (i.e. a total of 6 Wingate tests)*, whereas in the RL and RH trials, subjects will rest for the equivalent period of time (i.e. 30 min). For screening, potential subjects will come in the morning after an overnight fast. After obtaining informed consent, a series of screening tests will be conducted, including questionnaires (general health, physical activity and eating behaviour), anthropometry (height, weight, waist and hip circumference), blood pressure, resting heart rate, fasting blood glucose, HbA1c and body composition by air displacement plethysmography (BodPod, Cosmed, Rome, Italy). Following enrolment, subjects will undergo assessment of resting metabolic rate (RMR) for 30 minutes using a ventilated hood system (Quark CPET, Cosmed, Rome, Italy). RMR will be multiplied by a factor of 1.5 to approximate total energy requirement for weight maintenance. This will allow for tailoring the caloric content of the test meals to each subject's energy requirements. Thereafter, subjects will eat a small standardized breakfast and they will perform a 30-min SIT session to get familiarized with the exercise and the equipment. The total time required for screening will be around 2 hours. After the screening, subjects will be provided with a food diary to record all food intake on Day 1 and an activity diary to record all activities on Days 1 and 2 of the actual study trials (see below). Although only sedentary subjects will be recruited (=60 min of moderate-intensity exercise weekly), they will also be instructed to refrain from any vigorous activities during the three days before each study trials and throughout its duration. On Visits 2 to 5 (four experimental trials, in random order): Each of the four study visits will last for approximately 12 hours (spanning over 3 days), during which the following will take place: On Day 1, subjects will come to the Lab at around 4:00 pm to have the continuous glucose monitoring system (CGMS) inserted. CGMS will be used to measure 24 hour blood glucose concentrations. The sensor records interstitial blood glucose concentrations every five minutes. This will involve the insertion of a small sensor under the skin in the abdomen, which will be carried out by using a device that produces minimal pain and discomfort. After insertion, the stabilizing and calibration procedures will take 2 hours after which the subjects will go home with a standardized dinner to eat at around 7:00pm. Subjects will have to refrain from eating after 10:30pm and return to the CNRC the following morning (Day 2).On Day 2, subjects will report to the lab at 8:15 am following an overnight fast for the first of the four study conditions. Upon arrival, an indwelling catheter will be inserted into the antecubital fossa or forearm vein of one arm and will be kept patent. Blood samples will be obtained after the insertion of the catheter at 8:30 am (time = -30 min). Between 8:30 am and 9:00 am, subjects will either rest for 30 minutes or perform the SIT bout which will start with 4 ½ minutes of low-resistance cycling followed by 30 seconds of maximum effort, repeated for a total of 6 times*. During the SIT, subjects' ratings of perceived exertion (RPE) will be measured periodically using the Borg scale. At 9:00 am, blood samples will be collected (time = 0 min), after which breakfast (low or high GI) will be provided. After finishing breakfast, at 9:15 am, blood samples will be collected every 10 minutes for the first half hour and every 30 minutes for the remaining 3 hours at 15, 25, 35, 45, 75, 105, 135, 165, and 195 minutes. Before lunch is served at 12:45pm (time = 225 min), blood will be collected and again after lunch at 1:00 pm (time = 240 min), followed by blood collection every 10 minutes for the first half hour and every 30 minutes for the remaining 3 hours at 250, 260, 270, 300, 330, 360, 390, 420 and 450 minutes. After the last blood sample is collected at 4:30 pm, the catheter will be removed and the subjects will be discharged from the Lab. Subjects will be provided with the last test meal of the day (dinner) to eat at home at around 7:00pm. Throughout the day and at specific times, subjects will complete computerized visual analogue scales (VAS) on hunger and fullness. Blood samples will be used to measure fasting and postprandial concentrations of glucose and major glucoregulatory hormones like insulin and glucagon. C-peptide concentrations will be used to provide estimates of insulin secretion with mathematical modelling. Blood lactate will be determined before and after exercise to verify maximal exercise effort. On Day 3, subjects will come to the Lab at 8:30 am for final calibration and removal of the CGMS sensor. Subjects will come to the Lab for visits 3, 4, and 5 to perform the other 3 experimental trials, with at least 3 days wash-out in-between visits.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 21-40 years
* Chinese Ethnicity
* Body mass index between 17 - 25 kg m2
* Fasting blood glucose (< 6 mmol/L)
* Normal blood pressure (< 140/90 mmHg)
* Do not have metabolic diseases (such as diabetes, hypertension etc.)
* Do not have glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Do not take prescription medication that may affect metabolism
* Low activity level (≤ 60 min of moderate-intensity exercise weekly)
* Do not intentionally restrict food intake
* Do not have intolerances or allergies to test foods

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male voluteers
Enrollment: 16 (Actual)
Dates: Start 2015-12-17; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | up to 24 hours
  Measured using continuous glucose monitoring system
Glycaemic response | up to 8 hours
  Venous blood obtained through cannula, analysed using COBAS Analyzer

SECONDARY OUTCOMES:
Blood biochemistry | up to 8 hours
  Measure of plasma insulin, triglyceride, C-peptide, non-esterified fatty acid (NEFA) and lactate.
Hunger and satiety | up to 8 hours
  Assessed using Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No